CLINICAL TRIAL: NCT04503538
Title: Telemedicine for Early Detection of Cytokine Release Syndrome and Neurotoxicity Following CAR-T Infusion on an Outpatient Basis
Brief Title: Telemedicine for Early Detection of Cytokine Release Syndrome and Neurotoxicity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator decided not to pursue trial
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00067341; WFBCCC 99520 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Large B-cell Lymphoma; Diffuse Large B Cell Lymphoma; Primary Mediastinal Large B Cell Lymphoma; High-grade B-cell Lymphoma; Follicular Lymphoma
Keywords: Relapsed large B-cell lymphoma; Refractory large B-cell lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cell therapy and Telemedicine (Other): All outpatient CAR-T patients will require assessments for cytokine release syndrome and neurotoxicity three times daily (every 8 hours)
  Interventions: Other: Telemedicine visit

INTERVENTIONS:
Other: Telemedicine visit — Participants will be provided with a Wifi-and cellular enabled electronic tablet. Additionally, participants will receive a kit that contains a thermometer, a blood pressure monitoring cuff, and a pulse oximeter (to measure oxygen saturation level). Participants will attend an educational session to learn how the telemedicine visit works. Caregivers should attend with participants and will be trained to take temperatures, blood pressures, and oxygen saturation levels. Participants will also be asked to complete a test telehealth visit.

SUMMARY:
The purpose of this research is to replace one of participants' outpatient chimeric antigen receptor T-cell (CAR-T) therapy follow up visits with a virtual or "telemedicine" visit. The telemedicine visit will use an electronic tablet with a camera and a microphone that allows participants to communicate with their physicians and nurses. Participants will be provided with the necessary equipment to complete these visits.

DETAILED DESCRIPTION:
Primary Objective: To determine feasibility of telemedicine for outpatient cytokine release syndrome and neurotoxicity assessment (how many telemedicine visits successfully completed per patient)

Secondary Objective(s)

* To determine how many times a telemedicine visit triggered an action (inpatient admission/ outpatient observation status)
* To determine how many patients were detected to have cytokine release syndrome and/or neurotoxicity based on their telemedicine visit

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed relapsed or refractory large B-cell lymphoma after two or more lines of systemic therapy, including diffuse large B-cell lymphoma (DLBCL) not otherwise specified, primary mediastinal large B-cell lymphoma, high grade B-cell lymphoma, and DLBCL arising from of follicular lymphoma
* Age ≥ 18 years
* ECOG or Karnofsky performance status of ≤ 2
* Patients must have a caregiver(s) with them 24 hours a day for the first 30 days after CAR-T cell infusion
* Patients must stay within a 30-minute distance from the cancer center
* Patients must have access to wifi network or a cellular network
* Patients and caregiver(s) participating in patient's care must attend the education session for outpatient CAR-T and demonstrate competency to collect vital signs with equipment provided
* Must have the ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria:

* Patients who have acute lymphoblastic leukemia/lymphoma
* Patients who have a high tumor burden (> 10 cm largest mass) have a high risk of CRS who will receive CAR-T as an inpatient
* Patient or caregiver unable to understand and follow English language
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Number of Successfully Completed Telemedicine Visits | 3 years
  To determine feasibility of telemedicine for outpatient cytokine release syndrome and neurotoxicity assessment. Investigators will consider telemedicine feasible in this population if at least 13 of the 15 patients successfully complete 80% of telemedicine visits. A visit will be considered successful if all measurements are recorded OR if the visit is interrupted because the participant needs to come into the CAR-T unit for assessment. If a patient is admitted, then the 80% benchmark will be calculated based on the number of days the patient was outpatient at 11 pm. The proportion meeting the 80% benchmark will be reported along with an exact 95% confidence interval.

SECONDARY OUTCOMES:
Number of Times a Telemedicine Visit Triggered Action | 3 years
  To determine how many times a telemedicine visit triggered an inpatient admission or outpatient observation status
Number of Patients to Have Cytokine Release Syndrome | 3 years
  Descriptive statistics will be used to characterize the number of cases of cytokine release syndrome based on telemedicine visits.
Number of Patients to Have Neurotoxicity | 3 years
  Descriptive statistics will be used to characterize the number neurotoxicities reported based on telemedicine visits.

CONTACTS AND LOCATIONS:
Overall Officials: Rakhee Vaidya, MBBS, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No